CLINICAL TRIAL: NCT04917133
Title: Effect of Adapted Physical Activity, During Rehabilitation Stay, on Abilities and Quality of Life of Huntington Patients and Their Relatives "HUNT'ACTIV-MH-REHAB MOVE MORE TO LIVE BETTER"
Brief Title: Adapted Physical Activity Effect on Abilities and Quality of Life of Huntington Patients and Relatives During Rehab Stay
Acronym: HUNT'ACTIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Euromov Digital Health in Motion Montpellier France (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: APHP210469; 2021-A00423-38 (Other: IDRCB)
Record Dates: First submitted 2021-05-10; First posted 2021-06-08 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2022-09

CONDITIONS: Huntington Disease
Keywords: Adapted Physical Activity; Huntington's disease; rehabilitation
MeSH Terms: conditions — Huntington Disease

STUDY DESIGN:
Intervention Model Description: controlled randomized trial with two parallel arms
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adapted Physical workshops (Experimental): The experimental APA group will have in addition of the classic program, 6 APA workshops per week with collective care : Adapted Physical workshops, adapted cycling, therapeutic (horseback/equestrian) riding, cultural or leisure outings, situation tests
  Interventions: Behavioral: Adapted Physical Activity program
- Control (Other): Standard of care The control group will have the "classic" program performed in the standard of care with : kinesitherapy, soft gym, medico-social workshop, cognitive workshop, creative workshop, individual care (rehabilitation, rest, creation).
  Interventions: Other: Control

INTERVENTIONS:
Behavioral: Adapted Physical Activity program — classic 4-week rehabilitation program (standard care) + 6 APA workshops per week with collective care
  Arms: Adapted Physical workshops
Other: Control — classic 4-week rehabilitation program (standard care)
  Arms: Control

SUMMARY:
Intro:

Huntington's disease is a neurodegenerative disease that affects the brain, inducing a dysfunction and death of the middle spiny striatal projection neurons and a progressive alteration of cognitive and motor functions, and psycho-behavioral problems. There is currently no curative treatment but we know hat a multidisciplinary care can optimize the functioning and the quality of life of the patients with Huntington's disease.

A meta-analysis of 18studies indicates that exercise and physical activity can improve motor function, gait speed and balance, and would also improve self-confidence, independence, well-being, reduced apathy and better socialization with family and friends.

Hypothesis/Objective The hypothesis is that the inclusion of a 4 week-program with Adapted Physical Activity (APA) during a rehabilitation stay will improve some motor, cognitive and psycho-behavioral abilities, compared to the control group.

Method

The patients will be randomized into two groups :

The control group will have the "classic" program performed in the standard of care with: kinesitherapy, soft gym, medico-social workshop, cognitive workshop, creative workshop, individual care (rehabilitation, rest, and creation).

The experimental APA group will have in addition of the classic program, 6 APA workshops per week with collective support : Adapted Physical workshops, adapted cycling, therapeutic (horseback/equestrian) riding, cultural or leisure outings, situation tests

For the two groups, at the start of the 4 weeks of rehabilitation program an initial visit will be performed with, as part of this research, a clinical examination, a neurological examination, a dietary consultation, as well as a biological assessment as part of habitual care.

The clinical examination, the neurological examination and the dietary consultation will be performed each week, during the 4 weeks of the program,

At the end of the study, one month after the rehabilitation of the patient, a visit by phone-call will be performed for the patient and his caregiver.

ELIGIBILITY:
Inclusion Criteria for the Patient :

* Mid-stage Huntington's disease but with the ability for an autonomous walking for 10 meter
* Age ≥ 18 years old
* Stable medication for at least 4 weeks before the start of the study and a stable diet during the duration of the program. A stable diet means no weight loss up to 2kg in the last month prior to inclusion
* Patient who received a complete information and who signed an informed consent for the research (or his/her caregiver if incapacity to sign). Tutor/Guardian who received a complete information and who signed an informed consent for the research if applicable
* Affiliated to a social security scheme

Inclusion Criteria for the Caregiver :

* Person participating in the daily life of the patient
* The patient is included in the research
* Age ≥ 18 years old
* Having received a complete information
* Non opposition collected by the investigator

Exclusion Criteria:

* Having a physical or psychiatric condition preventing the completion of the program and assessments.
* Having a history of additional major neurological disorders such as a stroke or an orthopedic condition limiting mobility
* Any difficulty to understand or read French which could possibly invalidate the relevance of the application of questionnaires according to the opinion of the investigator
* Addictions, alcohol dependence
* Any other neurological, musculoskeletal or cardiovascular disease which could lead to errors in the assessment
* Participation to another interventional research or being in the exclusion period following a previous research if applicable
* Patient under AME (except if exemption from affiliation)

Exclusion criteria for the Caregiver :

* Having a physical or psychiatric condition preventing the completion of the program and assessments.
* Any difficulty to understand or read French which could possibly invalidate the relevance of the application of questionnaires according to the opinion of the investigator
* Under tutelage or guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2021-06-07 (Actual); Primary Completion 2021-12-07 (Actual); Study Completion 2021-12-07 (Actual)

PRIMARY OUTCOMES:
Motor function score of Unified Huntington's Disease Rating Scale (UHDRS) | Change from Baseline at 1 month
  UHDRS:Unified Huntington's Disease Rating Scale , minimum value: 0 maximum value: 124 higher score means a worse outcome Success will be defined by an improvement of the motor function score

SECONDARY OUTCOMES:
cognitive function score of Unified Huntington's Disease Rating Scale (UHDRS) using Stroop test | Change from Baseline at 1 month
  UHDRS:Unified Huntington's Disease Rating Scale , minimal number of correct answers:0 maximal number of correct answers:100 higher score means a better outcome Success will be defined by an improvement of the cognitive function score
psycho-behavioral function score of Unified Huntington's Disease Rating Scale (UHDRS) | Change from Baseline at 1 month
  UHDRS:Unified Huntington's Disease Rating Scale , minimum value:0 maximal value:88 higher score means a worse outcome Success will be defined by an improvement of the behavioral function score

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-André Natella, PhD, Study Director — Assistance Publique - Hôpitaux Paris
Locations (1):
- Hôpital Marin de Hendaye, Hendaye, France

IPD SHARING:
Plan to Share IPD: No
APHP IS DATA'S OWNER, PLEASE CONTACT BOARD